CLINICAL TRIAL: NCT04831177
Title: Thin-Flap Laser in Situ Keratomileusis Associated Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFLADE
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Myopic LASIK Candidates With Spherical Equivalent up to - 10 Diopters
Keywords: Dry eye; Femtolaser; Laser in situ keratomileusis
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients planned to undergo Femtosecond laser FS assisted LASIK (Active Comparator): In FS group, Allegretto WaveLight FS-200 femtosecond laser was used to create flaps with flap thickness planned to be 100 um.
  Interventions: Procedure: Laser in situ keratomileusis
- Patients planned to undergo Microkeratome MK assisted LASIK (Active Comparator): In MK group, Moria 2 Microkeratome was used to create flaps with flap thickness planned to be 100 um.
  Interventions: Procedure: Laser in situ keratomileusis

INTERVENTIONS:
Procedure: Laser in situ keratomileusis — Laser in situ keratomileusis LASIK is a procedure used to correct different types of ametropia through a creation of corneal flap whether with femtosecond laser or mechanically with a microkeratome followed by application of excimer laser to correct different refractive errors including Myopia, Hyperopia and Astigmatism.

SUMMARY:
Laser in situ keratomileusis (LASIK) eye surgery continues to be the most common refractive procedure used to correct different forms of ametropia. Although the introduction of femtosecond technology has markedly reduced the incidence of intraoperative flap complications and allowed a better control on flap parameters, dry eye remains one of the most challenging postoperative complications.

DETAILED DESCRIPTION:
The pathophysiology of post LASIK dry eye is not clear; however, many mechanisms have been suggested including inflammation, loss of conjunctival goblet cells during suction, exacerbation of a preexisting dry eye, abnormal interaction between the lid margins and the ocular surface. Intact corneal sensation is crucial for proper tear production and distribution on the ocular surface as well as maintaining the normal dynamics of eyelid blinking. Disruption of corneal nerves in LASIK decreases the release of neurotrophic factors necessary for the normal function of the corneal epithelium as well as the integrity of the lacrimal functional unit, a condition referred to as LASIK induced neurotrophic epitheliopathy (LINE) that largely contributes to the development of post- LASIK dry eye .

Many studies evaluated the incidence of post-refractive dry eye after LASIK compared to flapless laser vision correction (LVC) procedures such as PRK and small incision lenticule extraction (SMILE). The aim of this study is to assess and compare different dry eye parameters following LASIK with planned thin flaps created by femtosecond laser (FS) and mechanical microkeratome (MK).

ELIGIBILITY:
Inclusion Criteria:

1. Candidates for Laser Vision Correction (LVC).
2. Eyes with spherical equivalent (SE) up to - 10 diopters (D),
3. Corneal thickness at thinnest location of ≥ 500 um and estimated postoperative residual stromal bed of at least 300 um

Exclusion Criteria:

1. Patients with symptoms or signs of dry eye (TBUT <10 sec, Schirmer I test <10mm and Ocular Surface Disease Index OSDI score >13),
2. Posterior blepharitis, contact lens wearers ,
3. Ocular surface disease ,
4. Systemic diseases contraindicating LASIK and previous ocular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Tear film break up time TBUT | 6 months
  Fluorescein strip was inserted in the lower conjunctival fornix for few seconds then removed and the patient was asked to frequently blink, the stained tear film was observed with slit lamp (cobalt blue filter) till the appearance of the first black (dry) spot and the time interval in seconds was measured
Schirmer I test | 6 months
  Whatman filter paper (35 mm long) was folded 5mm and inserted in the lower conjunctival fornix away from the cornea and the patient was asked to blink normally. After 5minutes the paper was removed, and the amount of wetting in millimeters was measured.
Ocular Surface Disease Index OSDI | 6 months
  A questionnaire consisting of 12 questions. Each question with a score from 0 to 4, the OSDI score is calculated by multiplying the sum by 25 and dividing by the number of questions answered. This yields a score from 0 to 100. The results of OSDI score can be graded as normal (0-12), mild dry eye (13-22), moderate dry eye (23-32), or severe dry eye (33-100)
Lower Tear meniscus height (LTMH) | 6 months
  Anterior segment Optical coherence tomography (AS-OCT) examination was scheduled in the afternoon. The lower TMH was evaluated with a vertical scan centered on the inferior cornea and the lower eyelid. The lower TMH was measured with a special caliper tool incorporated in the device in micrometers and the height of the tear meniscus is the distance between 2 points ,one where the meniscus intersects the inferior cornea superiorly and the other where the meniscus intersects the lower eyelid margin inferiorly.
Lower Tear meniscus area (LTMA) | 6 months
  The lower TMA was evaluated using AS-OCT with a vertical scan centered on the inferior cornea and the lower eyelid then a built in software caliper tool was used to determine the borders of the tear meniscus and calculate the area (TMA) in millimeter square (mm2).

CONTACTS AND LOCATIONS:
Locations (1):
- TIBA eye center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sambhi RS, Sambhi GDS, Mather R, Malvankar-Mehta MS. Dry eye after refractive surgery: a meta-analysis. Can J Ophthalmol. 2020 Apr;55(2):99-106. doi: 10.1016/j.jcjo.2019.07.005. Epub 2019 Aug 20. PMID 31712000